CLINICAL TRIAL: NCT06813742
Title: A Prospective Exploratory Study Evaluating the Diagnostic Usefulness of 18F-mFBG PET Imaging in Pheochromocytoma
Brief Title: 18F-mFBG PET Imaging in the Evaluation of Pheochromocytoma
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: FAHZU-MFBG-PHEO
Record Dates: First submitted 2024-12-24; First posted 2025-02-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2024-12

CONDITIONS: Pheochromocytoma
MeSH Terms: conditions — Pheochromocytoma | interventions — 3-fluorobenzylguanidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 18F-MFBG PET/CT in Pheochromocytoma: Each patient receive a single intravenous injection of 18F-MFBG 5.55 MBq/kg and undergo PET/CT or PET/MR scan after 60 min post-injection.
  Interventions: Drug: 18F-MFBG

INTERVENTIONS:
Drug: 18F-MFBG — Patients with pheochromocytoma malignancies receive 5.55 MBq/kg of 18F-MFBG intravenously followed by PET/CT or PET/MR after 60min of injection.

SUMMARY:
The aim of this study is to evaluate the diagnostic performance and tumor burden of 18F-metafluorobenzylguanidine (18F-MFBG) positron emission tomography (PET) in patients with pheochromocytoma.

DETAILED DESCRIPTION:
Pheochromocytoma highly expresses norepinephrine transporter (NET) which is targeted by function alanalogue of norepinephrine, 123/131I-MlBG. However, low spatial resolution of 123/131I-MlBG and inaccurate attenuation correction of single photon emission tomography (SPECT/CT) will affect the image quality of MlBG SPECT and lead to poor diagnosis of small lesions. In addition, 123l-MlBG imaging is usually performed at 24h after injection, while 131I-MlBG is performed at 48h or even 72h after injection. The procedure is complicated and takes a long time, which limits clinical application. 18F-labeled MFBG is an ideal tracer to show the expression of NET. Preliminary data show that 18F-MFBG imaging is safe and has favorable biodistribution and kinetics with good targeting of lesions. Patients can undergo PET 0.5 hours after injection without special preparation. Our study will assess the safety profile, image quality and evaluate the diagnostic performance and tumor burden of 18F-MFBG. Patients with suspected or histologically confirmed pheochromocytoma will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 30-80 years old, primary school or above, with a regular caregiver;
2. Clinically diagnosed patients with pheochromocytoma;
3. Can provide informed consent, can understand and comply with the study requirements.

Exclusion Criteria:

1. Patients with serious primary diseases such as heart, brain, liver, kidney and hematopoietic system;
2. Uncontrolled hypertension or high-risk BP (i.e., systolic BP > 180 mmHg or diastolic BP > 110 mmHg);
3. Patients with mental disorders or primary affective disorders;
4. Unable to understand and adhere to the study protocol or provide informed consent;
5. Contraindications to PET imaging (including pregnant women, lactating women, and women of childbearing age with recent childbearing plans, etc.);
6. Allergy to imaging agents;
7. Patients who were unable to cooperate with PET scanning, such as hypoglycemia, severe pain or tremor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with suspected or confirmed pheochromocytoma
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between positive and negative 18F-mFBG PET/CT or PET/MR Imaging and pathological diagnosis and treatment effect in patients with pheochromocytoma. | through study completion, an average of 1 year
  Main outcome measure

SECONDARY OUTCOMES:
False positive and false negative results of 18F-mFBG PET/CT or PET/MR Imaging in patients with pheochromocytoma. | through study completion, an average of 1 year
  Secondary outcome measure

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang